CLINICAL TRIAL: NCT02820220
Title: Knowledge and Perceptions Regarding Janani Shishu Suraksha Karyakram (JSSK) and Rashtriya Bal Swasthya Karyakram (RBSK) Programs in the Patients/Patient Attendants,Nursing Students and in Service Nurses: A Comparative Study
Brief Title: Knowledge and Perceptions Regarding JSSK and RBSK in Patients and Nurses: A Comparative Study
Status: Completed | Type: Observational
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, DR. VIKRAM DATTA, Principal Investigator, Lady Hardinge Medical College
Other Study IDs: LadyHardingeMC
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Knowledge Maternal-Child Health Services
Keywords: Knowledge; Programs; Patients; Students; Nurses

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patient/patient attendants: 1. Study subjects will be females.
  2. Age at enrolment should be more than 18 years.
  3. Attending Department of Paediatrics OPD/emergency/well-baby clinics/immunisation clinics OR Department of Gynaecology and Obstetrics OPD/emergency/Ante-natal clinics/Post-natal clinics of Lady Hardinge Medical College and associated hospitals.
  4. Written informed consent to participate in the study.
- Students,nursing: 1. Pursuing Bsc Nursing(in their final year) or intern of college of nursing LHMC
  2. Written informed consent to participate in the study
- In-service nurses: 1. Posted in Department of Paediatrics indoor/OPD/well-baby clinics/immunisation clinics or Department of Gynaecology and Obstetrics indoor/OPD/emergency/Ante-natal clinics/Post-natal clinics of Lady Hardinge Medical College and associated hospitals.
  2. Written informed consent to participate in the study.

SUMMARY:
Observational, cross sectional study, carried out with the help of a pre-designed and pre-tested questionnaire with the research hypothesis as: Knowledge and perception regarding JSSK and RBSK in nursing students is better as compared to in-service nurses as well as patients/patient attendants (attending LHMC and associated hospitals, New Delhi, India)

DETAILED DESCRIPTION:
The objectives of the study were to:

1. To study knowledge and perceptions regarding JSSK and RBSK programs in the patients/patient attendants, nursing students and in-service nurses attending LHMC and associated hospitals.
2. To compare knowledge and perceptions regarding JSSK and RBSK programs in the patients/patient attendants, nursing students and in-service nurses attending LHMC and associated hospitals.
3. To identify factors contributing to knowledge regarding JSSK and RBSK programs in the patients/patient attendants, nursing students and in-service nurses attending LHMC and associated hospitals.

ELIGIBILITY:
Inclusion Criteria:

Group 1) Patients/Attendants:

* All study subjects must be female.
* Age more than 18 years.
* Written informed consent to participate in the study.

Group 2) Nursing Student:

* Students / intern at College of nursing LHMC pursuing Bsc Nursing
* Written informed consent to participate in the study

Group 3) In-service Nurses:

* Posted in Department of Paediatrics indoor/OPD/well-baby clinics/immunisation clinics or Department of Gynaecology and Obstetrics indoor/OPD/emergency/Ante-natal clinics/Post-natal clinics of Lady Hardinge Medical College and associated hospitals.
* Written informed consent to participate in the study

Exclusion Criteria:

* Males for the patient/attendant group 1

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 participants enrolled from the patients/attendant subset,93 Nursing students(final year) and interns from the Nursing college, LHMC along with 100 nurses posted in the LHMC and associated hospitals enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Knowledge and perception regarding JSSK and RBSK in study population groups | 90 days
  The knowledge and perception will be evaluated by yes, no responses using predesigned and pretested questionnaire presented to each of the three study groups.

SECONDARY OUTCOMES:
Comparison of the knowledge and perception regarding JSSK and RBSK in study population groups | 90 days
  The knowledge and perception will be compared using yes and no responses obtained on predesigned and pretested questionnaire presented to each of the three study groups.
Study of factors contributing to knowledge regarding JSSK and RBSK in study population groups | 90 days
  The factors will be identified and evaluated using yes and no responses obtained on the predesigned and pretested questionnaire presented to each of the three study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Datta, MD,DNB, Study Chair — Lady Hardinge Medical College,New Delhi,India

IPD SHARING:
Plan to Share IPD: Undecided